CLINICAL TRIAL: NCT05605340
Title: Use of Home-delivered Meals to Reduce Excessive Gestational Weight Gain for High-risk Women
Brief Title: Healthier At-home Meals for Expectant Mothers
Acronym: Her HOME
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Gareth R. Dutton PhD, Primary Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-300009275; R21HD107325 (NIH)
Record Dates: First submitted 2022-10-25; First posted 2022-11-04 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Pregnancy Related; Weight Gain, Maternal
Keywords: Maternal Overweight; Maternal Obesity; Gestational weight gain; Meal delivery
MeSH Terms: conditions — Gestational Weight Gain; Pregnancy in Obesity

STUDY DESIGN:
Intervention Model Description: All participants enrolled will receive the study intervention. A quasi-experimental design will be used to investigate the preliminary efficacy of the meal delivery intervention on gestational weight gain and estimate the effect size of the intervention relative to a non-randomized standard care but weighted control group derived from de-identified hospital records.
Masking Description: All participants enrolled will receive the study intervention, so blinding is not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Meal delivery intervention with brief behavioral support.
  Interventions: Behavioral: Meal Delivery

INTERVENTIONS:
Behavioral: Meal Delivery — 10 healthy, home-delivered meals per week + brief weekly remote behavioral support

SUMMARY:
This study is being done to test the feasibility, acceptability, and preliminary efficacy of a meal delivery intervention for managing gestational weight gain among pregnant women with overweight or obesity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Gestational age ≤ 15 weeks as assessed by ultrasound
* Body mass index (BMI) ≥ 25 kg/m2
* Singleton viable pregnancy
* Receiving care and planning to deliver at UAB
* Residing within the delivery radius of the meal delivery company
* Wi-Fi or Bluetooth Internet connection in home (for digital Wi-Fi enabled study scale)

Exclusion Criteria:

* Self-reported major health conditions (e.g., heart disease, cancer, renal disease, and Type 1 or Type 2 diabetes)
* Current substance abuse
* Current treatment for serious psychiatric disorder (schizophrenia, bipolar disorder)
* Known fetal anomaly
* Planned termination of pregnancy
* Past history or current diagnosis of anorexia or bulimia
* Current use of one or more of the following medications:
* Metformin
* Systemic steroids
* Antipsychotic agents
* Anti-seizure medications or mood stabilizers that would be expected to have a significant impact on body weight
* Medications for ADHD including amphetamines and methylphenidate
* Any teratogenic agent Class D
* Participation in another dietary and/or weight management intervention during pregnancy
* Unwilling or unable to consume prepared meals delivered weekly
* Unable to understand and communicate in verbal and written English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-08-09 (Actual); Primary Completion 2025-10-14 (Actual); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in weight from first to last prenatal visit | First prenatal visit (<15 weeks gestation), last prenatal visit (35+ weeks gestation)
  Weight measured at each prenatal visit will be retrieved from medical records for all participants and used to model total weight change from the first to the last prenatal visit (i.e., gestational weight gain).

SECONDARY OUTCOMES:
Change in Food Insecurity | baseline (12-15 weeks gestation), (35-36 weeks gestation)
  Determined using the 18-item United States (US) Household Food Security Survey Module based on the previous 30 days. Adult food security scores range from 0 to 10, with lower values indicating greater food security.
Change in Perceived Stress | baseline (12-15 weeks gestation), (35-36 weeks gestation)
  Determined using the 10-item Perceived Stress Scale (PSS-10) based on the last month. PSS-10 scores range from 0 to 40, with higher scores representing higher levels of perceived stress.
Change in Participant Satisfaction with Diet | baseline (12-15 weeks gestation), (35-36 weeks gestation)
  Determined using the 28-item Diet Satisfaction Questionnaire in which participants respond to 28 statements using a 5-point Likert scale. Responses are average to produce a total diet satisfaction score ranging from 1-5. Changes in overall diet satisfaction, as well as changes in subscale scores for Cost Factor and Planning & Preparation Factor will be examined from baseline to follow-up.
Proportion of Women Exceeding Institute of Medicine Gestational Weight Gain Guidelines | First prenatal visit (<15 weeks gestation), last prenatal visit (35+ weeks gestation)
  Weight at the first prenatal visit will be subtracted from weight at the last prenatal visit. Women will be categorized as exceeding 2009 Institute of Medicine gestational weight gain guidelines if the difference is > 11.5 kg gain for women with overweight or >9 kg for women with obesity at the first prenatal visit.

CONTACTS AND LOCATIONS:
Overall Officials: Gareth Dutton, PhD, Principal Investigator — University of Alabama at Birmingham; Camille Worthington, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in a publication will be made available upon request beginning 9 months and ending 36 months following article publication. The research team will keep a record of all individuals and/or research teams who request and receive a copy of the project data. Interested investigators will be asked to submit a document indicating the specific aims of the analyses, the analytic plan, available resources for completing the proposed project, proposed timeline, and goals (i.e., manuscripts, presentations, and/or grant applications). The PI and research team will review these requests to determine whether the proposed analyses constitute an innovative and significant exploration of the data, whether the proposed team has sufficient resources to complete the request, and whether data will be adequately protected and managed.
Supporting Information: Study Protocol, ICF
Time Frame: Data requests can be submitted starting 9 months after publication of results and ending 36 months following article publication.
Access Criteria: Access to IPD stripped of all HIPAA identifiers (except age) for this study can be requested by qualified researchers engaging in independent scientific research whose proposed research has received Institutional Review Board approval, and will be provided following review and approval of a research proposal and timeline, statistical analysis plan, and goals (e.g., manuscripts, presentations, grant applications). The Principal Investigator (PI) and research team will review these requests to determine whether the proposed analyses constitute an innovative and significant exploration of the data, whether the proposed team has sufficient resources to complete the request, and whether data will be adequately protected and managed. Based on institutional policies, execution of a Data Sharing Agreement may be required prior to sharing of IPD. IPD requests can be made to the MPIs at gdutton@uabmc.edu or cschneid@uab.edu.